CLINICAL TRIAL: NCT03896217
Title: A Double-blind, Randomised, Placebo-controlled Single-site Study of High Dose Simvastatin Treatment for Secondary Progressive Multiple Sclerosis: Impact on Vascular Perfusion and Oxidative Damage
Brief Title: Simvastatin in Secondary Progressive Multiple Sclerosis
Acronym: MS-OPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/0730 & 2017-003008-30
Record Dates: First submitted 2018-10-26; First posted 2019-03-29 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: Multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simvastatin (Active Comparator): Simvastatin is part of the pharmacotherapeutic group of HMG-CoA reductase inhibitors (ATC-Code: C10A A01). Simvastatin is licensed within the EU for hypercholesterolemia and cardiovascular prevention but for this trial its use will be outside its licensed indication. Oral Simvastatin will be taken 40mg daily (one tablet in the evening) for 4 weeks and then at week 4 up titrated to 80mg daily (two tablets in the evening.
  Interventions: Drug: Simvastatin
- Placebo (Placebo Comparator): Matched Placebo (one tablet in the evening) for 4 weeks and then at week 4 up titrated to two tablets daily in the evening.
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Simvastatin — Simvastatin 40mg for first 4 weeks and 80mg (if tolerated) thereafter up to 17 weeks
  Other Names: ATC-Code: C10A A01

SUMMARY:
Multiple sclerosis (MS) is a neurological condition which is a common cause of disability in young people. It is thought to be an autoimmune condition, where the body's immune system begins to attack itself. The cause of MS is unknown but is thought to be a mix of genetic and environmental factors. There are treatments available for early stages of MS, but the later stage known as Secondary Progressive MS (SPMS) has no current treatment.

Statins are a safe treatment traditionally used to reduce cholesterol levels. However, statins also have other effects which could reduce the progression of SPMS, such as effects on the immune system and circulation. A recent study (Chataway et al., 2014) showed that treatment with high-dose simvastatin, a type of statin, reduced the progression of SPMS but no effect on the immune system was seen. It is possible that simvastatin does not treat the immune system but improves how the blood and blood vessels in the brain work in this disease.

The purpose of the clinical trial is to test how Simvastatin (80mg/day) may slow down disease progression in people living with SPMS compared to placebo (dummy pill). Participants will receive either Simvastatin or placebo and will be asked to take 2 tablets daily, for up to 17 weeks.

DETAILED DESCRIPTION:
Approximately 60% of those affected with relapsing-remitting MS (RRMS) enter a SPMS stage after a median interval of 10 to 15 years, where disability accumulates gradually in the absence of relapses. A smaller proportion (15%), run a progressive course from onset (primary progressive (PP) MS). The progressive, "neurodegenerative" component of MS, rather than the clinical deficit resulting from incomplete recovery from each relapse in RRMS, is the dominant cause of long-term disability. Whilst over ten therapies are now licensed for RRMS, no treatment strategies, with the exception of a recent study by the investigators, have succeeded in slowing the progression of this later debilitating stage.

Optic neuritis, inflammation of the optic nerve, is a common event associated with MS resulting in 27% of subjects with residual visual impairment. The impact of damage arising from an inflammatory lesion in the optic nerve can be visualised using optical coherence tomography (OCT) as a reduction in both ganglion cell layer and retinal nerve fibre layer thickness. However it is increasingly being appreciated that a number of other inflammatory and neurodegenerative changes occur in the retina of MS patients. These retinal changes, reflecting both the disease and its level of activity, have highlighted its potential as a surrogate outcome measure to study preservation of neuronal and/or vascular structure/function after an inflammatory event or as the disease progresses.

During the last two decades there have been significant advances in the understanding of MS leading to treatment for the RRMS phase. Despite this, there has been a failure to find an effective treatment for progression and this remains a major unmet need, as highlighted by the International Progressive MS Alliance. The many challenges of progressive studies including optimal design, sensitive outcomes, suitable length and subject numbers are gradually being overcome by the MS community, but as yet extending the anti-inflammatory approach that has been effective in RRMS has not borne fruit in SPMS. Indeed the failure of the recent PPMS trial using fingolimod makes the success of simvastatin in the SPMS study all the more exciting, especially as the extensive systemic immunological assessment in this latter study revealed no impact on immune status. The real success of this simvastatin phase II study may be that it initiates novel avenues of investigation driven by the wide-ranging and well-characterised effects statins have on the body as well as a prelude to a definitive phase III trial. This premise underpins the research strategy.

Preclinical work has focused on the role played by the vascular barriers (the blood-brain and blood retinal barriers) in the inflammatory process and in particular how they support leukocyte traffic to the central nervous system (CNS). This research, along with that of others, led to the identification and characterisation of endothelial cell (EC) signalling processes that facilitate leukocyte diapedesis and activate pro-inflammatory responses. The investigators found that a key central regulator of the EC signalling pathway supporting leukocyte diapedesis was the small GTPase Rho, and this led to investigating whether small GTPases could be targeted pharmacologically to reduce aberrant leukocyte migration into the brain and retina. Since small GTPases require posttranslational lipid modification (prenylation) to become functional, the investigators tested whether inhibition of Rho prenylation with prenyl transferase inhibitors (PTIs) affects lymphocyte migration. Treatment of brain endothelial cell monolayers in vitro, or animals induced for experimental autoimmune encephalomyelitis (EAE, the animal model of MS), resulted in inhibition of lymphocyte migration and attenuation of the disease respectively.

Since the isoprenoids used for post-translational prenylation of small GTPases are derived from the cholesterol synthesis pathway, the investigators next investigated whether HMGCoA reductase inhibitors (statins) were also able to significantly inhibit Rho activity and reduce the severity of brain and retinal inflammatory disease. This research revealed that statins effectively reduced Rho prenylation and attenuated disease in experimentally induced models of MS and posterior uveitis. Whilst the investigators were able to demonstrate that one of the effects of statin treatment was to modify endothelia cell function and inhibit transendothelial migration of leukocytes, it is clear from many other experimental studies that efficacy may also be due to effects on other cell types such as immune cells.

Indeed, it is now widely recognised that statins have anti-inflammatory properties that operate independently of their cholesterol lowering effect. Accordingly, statins have been shown to inhibit MHC class II restricted Ag presentation, attenuate antigen-presenting cell maturation and down-regulate T cell activation and proliferation. Of those T cells that proliferate, statins induce a shift from a proinflammatory Th1 to a regulatory Th2 phenotype. In addition, statins block adhesion molecule expression and their interactions, inhibit the production of chemokines and their receptors, and reduce the secretion of matrix metalloproteinases. Activation of the transcription factor NFκB, an important activator of pro-inflammatory mediators, is also inhibited by statins, alongside a concomitant upregulation of endothelial cell protective genes. Finally, it has been shown that endothelial nitric oxide synthase (eNOS) activity is enhanced, whilst inducible NOS (iNOS) is inhibited.

This remarkable pleiotropic capacity for modulating the immune system and inflammation has prompted the clinical testing of statins for the treatment of RRMS and other inflammatory diseases. In one such study in 30 patients with RRMS, simvastatin (80mg) taken over 6 months reduced the number of brain lesions by 40%, although no change in disability scores was observed over this short study period. Other studies, however, have failed to demonstrate any significant clinical improvement in RRMS following statin treatment alone or in combination with other disease modifying drugs. Nevertheless, it should be noted that none of the studies so far have been sufficiently powered, rendering definitive conclusions impossible.

Whilst there is a clear-cut rationale for using statins for the treatment of RRMS, in SPMS there is less obvious justification, as disease progression in the absence of new plaque formation is thought to be due predominantly to neurodegeneration (or neuronal loss). This results from several mechanisms, including microglia activation, chronic oxidative injury, accumulation of mitochondrial damage in axons, and age-related iron accumulation in the human brain. Whereas large scale inflammatory lesions rarely occur at this stage of the disease, inflammation is prominent in progressive MS, where it is found throughout the grey and white matter, and in the meninges, with its most severe form being represented by the ectopic follicles that contribute to grey matter damage. This suggested that given their Immunomodulatory / anti-inflammatory actions, statins might still provide some benefit in SPMS. Nonetheless, neuronal loss is regarded as the key pathological feature, which raised the question whether statins also possess neuroprotective properties. Several lines of evidence suggest this may be the case.

Firstly, statins are increasingly seen as vasculoprotective with a capacity to improve vascular perfusion and maintain/enhance blood vessel function thus protecting against long-term chronic hypoxic damage. This is germane given the growing evidence that dysfunctional/reduced blood flow in MS may predispose the tissue to damage resulting in neuronal cell dysfunction and ultimately cell death. Such beneficial effects on microvascular perfusion may be mediated through statins enhancing eNOS activation and inhibiting endothelin-1.

Secondly, there are reports that statins may also be neuroprotective through reducing free radical damage either by improving blood flow and reducing hypoxia-mediated reactive oxygen species (ROS) production, or through direct inhibition of cytotoxic pathways. In the latter case, statins may protect neuroparenchymal cells via inhibition of iNOS in activated microglia and astrocytes, resulting in attenuated cytotoxic damage to neurons and oligodendrocytes. Furthermore, statins may also exert a neuroprotective effect by preventing glutamate-mediated excitotoxicity.

Together these data provided a compelling rationale for testing the potential therapeutic effect of statins in SPMS. In 2008, the investigators therefore embarked on a two-year double-blind, controlled trial of 140 patients, randomising them to either 80mg of simvastatin or placebo. The recently published results of this trial showed that brain atrophy was reduced by over 40% alongside a similar favourable effect on two major disability outcome measures. This is the first evidence of a drug having a beneficial effect on SPMS disease progression. Surprisingly, however, and contrary to expectations, the investigators did not identify any modulation of the immune system, raising the critical question of the mechanism of statin action.

It is the hypothesis, therefore, that the neuroprotective effects of statins in SPMS are mediated by stimulating enhanced microvascular perfusion and/or by inhibition of oxidative damage/neurotoxicity. This study will test this hypothesis.

There are no current treatments for SPMS. Given the investigators demonstrated that simvastatin was beneficial in a phase II trial but were unable to elucidate any mechanism, it is important to try and understand the mechanism of action to develop further therapies.

The investigators will investigate the impact of high dose simvastatin (80mg/day) on cerebral and retinal blood perfusion and vascular structure/function, brain neuroaxonal density and glutamate excitotoxicity in SPMS. In addition, various systemic parameters will be evaluated to determine the effect of high dose statin treatment on immune function, oxidative damage and vascular barrier function.

Simvastatin is being used outside of its posology and method of administration. The previous phase two trial found simvastatin was safe up to the maximum dose of 80 mg/day given as a single dose in the evening. Based on the recommendations of the SPC and previous studies, the proposed use of 80mg of Simvastatin will, therefore, be used for this study.

ELIGIBILITY:
Inclusion criteria:

1. Patients must have a confirmed diagnosis of multiple sclerosis according to revised Mc Donald criteria and have entered the secondary progressive stage or a diagnosis of Primary Progressive MS.(Polman et al., 2011, Lublin, 2014) Steady progression rather than relapse must be the major cause of increasing disability in the preceding 2 years. Progression can be evident from either an increase of at least one point on the EDSS or clinical documentation of increasing disability.
2. EDSS 4.0 - 6.5 (inclusive).
3. Male and Females aged 18 with no upper age limit
4. Females of childbearing potential and males with partners who are of childbearing age must be willing to use an effective method of contraception (Double barrier method of birth control or True abstinence) from the time consent is signed until 6 weeks after treatment discontinuation and inform the trial team if pregnancy occurs.

   For the purpose of clarity, True abstinence is when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence, withdrawal, spermicides only or lactational amenorrhoea method for the duration of a trial, are not acceptable methods of contraception.
5. Females of childbearing potential have a negative pregnancy test within 7 days prior to being registered/randomised. Participants are considered not of child bearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
6. Willing and able to comply with the trial protocol (e.g. can tolerate MRI and fulfils the requirements for MRI, e.g. not fitted with pacemakers or permanent hearing aids) ability to understand and complete questionnaires.
7. Willing and able to provide written informed consent.
8. Willing to ingest gelatine (placebo will contain this). Participants must therefore be informed sensitive to personal beliefs e.g. faith, diet.

Exclusion criteria:

1. Unable to give informed consent.
2. Those that have experienced a relapse or have been treated with steroids (both i.v. and oral) for multiple sclerosis relapse within 3 months of the screening visit.

   These patients may undergo a further screening visit once the 3 month window has expired and may be included if no steroid treatment has been administered in the intervening period. Patients on steroids for another medical condition may enter as long as the steroid prescription is not for multiple sclerosis (relapse/ progression).
3. Patient is already taking or is anticipated to be taking a statin or lomitapide for cholesterol control.
4. Any medications that unfavourably interact with statins as per Spc recommendations e.g.: fibrates, nicotinic acid, cyclosporin, azole anti-fungal preparations, macrolideantibiotics, protease inhibitors, nefazodone, verapamil, amiodarone, large amounts of grapefruit juice or alcohol abuse within 6 months.
5. The use of immunosuppressants (e.g. azathioprine, methotrexate, cyclosporin) or disease modifying treatments (avonex, rebif, betaferon, glatiramer, dimethyl fumerate, fingolimod) within the previous 6 months.
6. The use of mitoxantrone if treated within the last 12 months.
7. Patient has received treatment with alemtuzumab.
8. Use of other experimental disease modifying treatment (including research in an investigational medicinal product) within 6 months of baseline visit.
9. Active Hepatic disease or known severe renal failure (creatinine clearance <30ml/min).
10. Screening levels of alanine aminotransferase (ALT), aspartate aminotransferase (AST) or creatine kinase (CK) are three times the upper limit of normal patients.
11. If the patient reports any ophthalmic conditions such as glaucoma, ocular trauma or degenerative eye disease. . Cataracts are acceptable as long as they have not been advised to have surgery. No restrictions on post surgical care, unless the patient reports sight restricting capsule opacity. Short title: Simvastatin in Progressive MS Sponsor code: 16/0730 UCL protocol Version 1.7, dated 18/10/2022 Page 40 of 86
12. Patient unable to tolerate or unsuitable to have baseline MRI scan (e.g. metal implants, heart pacemaker) or MRI scan not of adequate quality for analysis (e.g.

    too much movement artefact).
13. Females who are pregnant, planning pregnancy or breastfeeding.
14. Allergies to IMP active substance or to any excipients of IMP and placebo or other conditions that contraindicate use of galactose (eg. Hereditary galactose intolerance, Lactase deficiency, glucose-galactose malabsorption)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2023-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Nicholas, MD, Principal Investigator — UCL
Locations (1):
- Department of Neuroinflammation, UCL Institute of Neurology, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No identifiable patient information will be supplied to other researchers external to the organisation.

REFERENCES:
- [Background] Chataway J, Schuerer N, Alsanousi A, Chan D, MacManus D, Hunter K, Anderson V, Bangham CR, Clegg S, Nielsen C, Fox NC, Wilkie D, Nicholas JM, Calder VL, Greenwood J, Frost C, Nicholas R. Effect of high-dose simvastatin on brain atrophy and disability in secondary progressive multiple sclerosis (MS-STAT): a randomised, placebo-controlled, phase 2 trial. Lancet. 2014 Jun 28;383(9936):2213-21. doi: 10.1016/S0140-6736(13)62242-4. Epub 2014 Mar 19. PMID 24655729
- [Background] Grecescu M. Optical coherence tomography versus visual evoked potentials in detecting subclinical visual impairment in multiple sclerosis. J Med Life. 2014 Oct-Dec;7(4):538-41. PMID 25713617
- [Background] Huang-Link YM, Al-Hawasi A, Lindehammar H. Acute optic neuritis: retinal ganglion cell loss precedes retinal nerve fiber thinning. Neurol Sci. 2015 Apr;36(4):617-20. doi: 10.1007/s10072-014-1982-3. Epub 2014 Oct 14. PMID 25311917
- [Background] Bennett JL, de Seze J, Lana-Peixoto M, Palace J, Waldman A, Schippling S, Tenembaum S, Banwell B, Greenberg B, Levy M, Fujihara K, Chan KH, Kim HJ, Asgari N, Sato DK, Saiz A, Wuerfel J, Zimmermann H, Green A, Villoslada P, Paul F; GJCF-ICC&BR. Neuromyelitis optica and multiple sclerosis: Seeing differences through optical coherence tomography. Mult Scler. 2015 May;21(6):678-88. doi: 10.1177/1352458514567216. Epub 2015 Feb 6. PMID 25662342
- [Background] Fox RJ, Thompson A, Baker D, Baneke P, Brown D, Browne P, Chandraratna D, Ciccarelli O, Coetzee T, Comi G, Feinstein A, Kapoor R, Lee K, Salvetti M, Sharrock K, Toosy A, Zaratin P, Zuidwijk K. Setting a research agenda for progressive multiple sclerosis: the International Collaborative on Progressive MS. Mult Scler. 2012 Nov;18(11):1534-40. doi: 10.1177/1352458512458169. Epub 2012 Aug 23. PMID 22917690
- [Background] Lublin F, Miller DH, Freedman MS, Cree BAC, Wolinsky JS, Weiner H, Lubetzki C, Hartung HP, Montalban X, Uitdehaag BMJ, Merschhemke M, Li B, Putzki N, Liu FC, Haring DA, Kappos L; INFORMS study investigators. Oral fingolimod in primary progressive multiple sclerosis (INFORMS): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet. 2016 Mar 12;387(10023):1075-1084. doi: 10.1016/S0140-6736(15)01314-8. Epub 2016 Jan 28. PMID 26827074
- [Background] Greenwood J, Heasman SJ, Alvarez JI, Prat A, Lyck R, Engelhardt B. Review: leucocyte-endothelial cell crosstalk at the blood-brain barrier: a prerequisite for successful immune cell entry to the brain. Neuropathol Appl Neurobiol. 2011 Feb;37(1):24-39. doi: 10.1111/j.1365-2990.2010.01140.x. PMID 20946472
- [Background] Walters CE, Pryce G, Hankey DJR, Sebti SM, Hamilton AD, Baker D, Greenwood J, Adamson P. Inhibition of Rho GTPases with protein prenyltransferase inhibitors prevents leukocyte recruitment to the central nervous system and attenuates clinical signs of disease in an animal model of multiple sclerosis. J Immunol. 2002 Apr 15;168(8):4087-4094. doi: 10.4049/jimmunol.168.8.4087. PMID 11937568
- [Background] Greenwood J, Walters CE, Pryce G, Kanuga N, Beraud E, Baker D, Adamson P. Lovastatin inhibits brain endothelial cell Rho-mediated lymphocyte migration and attenuates experimental autoimmune encephalomyelitis. FASEB J. 2003 May;17(8):905-7. doi: 10.1096/fj.02-1014fje. Epub 2003 Mar 5. PMID 12626426
- [Background] Harry R, Gegg M, Hankey D, Zambarakji H, Pryce G, Baker D, Calder V, Adamson P, Greenwood J. Suppression of autoimmune retinal disease by lovastatin does not require Th2 cytokine induction. J Immunol. 2005 Feb 15;174(4):2327-2335. doi: 10.4049/jimmunol.174.4.2327. PMID 15699169
- [Background] Greenwood J, Steinman L, Zamvil SS. Statin therapy and autoimmune disease: from protein prenylation to immunomodulation. Nat Rev Immunol. 2006 May;6(5):358-70. doi: 10.1038/nri1839. PMID 16639429
- [Background] Weber MS, Youssef S, Dunn SE, Prod'homme T, Neuhaus O, Stuve O, Greenwood J, Steinman L, Zamvil SS. Statins in the treatment of central nervous system autoimmune disease. J Neuroimmunol. 2006 Sep;178(1-2):140-8. doi: 10.1016/j.jneuroim.2006.06.006. Epub 2006 Jul 24. PMID 16860400
- [Background] Greenwood J, Mason JC. Statins and the vascular endothelial inflammatory response. Trends Immunol. 2007 Feb;28(2):88-98. doi: 10.1016/j.it.2006.12.003. Epub 2007 Jan 2. PMID 17197237
- [Background] Vollmer T, Key L, Durkalski V, Tyor W, Corboy J, Markovic-Plese S, Preiningerova J, Rizzo M, Singh I. Oral simvastatin treatment in relapsing-remitting multiple sclerosis. Lancet. 2004 May 15;363(9421):1607-8. doi: 10.1016/S0140-6736(04)16205-3. PMID 15145635
- [Background] Neuhaus O, Hartung HP. Evaluation of atorvastatin and simvastatin for treatment of multiple sclerosis. Expert Rev Neurother. 2007 May;7(5):547-56. doi: 10.1586/14737175.7.5.547. PMID 17492904
- [Background] Paraskevas KI. Statin treatment for rheumatoid arthritis: a promising novel indication. Clin Rheumatol. 2008 Mar;27(3):281-7. doi: 10.1007/s10067-007-0806-8. Epub 2007 Dec 8. PMID 18066611
- [Background] Yuan C, Zhou L, Cheng J, Zhang J, Teng Y, Huang M, Adcock IM, Barnes PJ, Yao X. Statins as potential therapeutic drug for asthma? Respir Res. 2012 Nov 24;13(1):108. doi: 10.1186/1465-9921-13-108. PMID 23176705
- [Background] Young RP, Hopkins RJ. Update on the potential role of statins in chronic obstructive pulmonary disease and its co-morbidities. Expert Rev Respir Med. 2013 Oct;7(5):533-44. doi: 10.1586/17476348.2013.838018. PMID 24138695
- [Background] Mahad DH, Trapp BD, Lassmann H. Pathological mechanisms in progressive multiple sclerosis. Lancet Neurol. 2015 Feb;14(2):183-93. doi: 10.1016/S1474-4422(14)70256-X. PMID 25772897
- [Background] Kutzelnigg A, Lucchinetti CF, Stadelmann C, Bruck W, Rauschka H, Bergmann M, Schmidbauer M, Parisi JE, Lassmann H. Cortical demyelination and diffuse white matter injury in multiple sclerosis. Brain. 2005 Nov;128(Pt 11):2705-12. doi: 10.1093/brain/awh641. Epub 2005 Oct 17. PMID 16230320
- [Background] Magliozzi R, Howell O, Vora A, Serafini B, Nicholas R, Puopolo M, Reynolds R, Aloisi F. Meningeal B-cell follicles in secondary progressive multiple sclerosis associate with early onset of disease and severe cortical pathology. Brain. 2007 Apr;130(Pt 4):1089-104. doi: 10.1093/brain/awm038. PMID 17438020
- [Background] Liao JK. Beyond lipid lowering: the role of statins in vascular protection. Int J Cardiol. 2002 Nov;86(1):5-18. doi: 10.1016/s0167-5273(02)00195-x. PMID 12243846
- [Background] Mason JC. Statins and their role in vascular protection. Clin Sci (Lond). 2003 Sep;105(3):251-66. doi: 10.1042/CS20030148. PMID 12793855
- [Background] Haendeler J, Hoffmann J, Zeiher AM, Dimmeler S. Antioxidant effects of statins via S-nitrosylation and activation of thioredoxin in endothelial cells: a novel vasculoprotective function of statins. Circulation. 2004 Aug 17;110(7):856-61. doi: 10.1161/01.CIR.0000138743.09012.93. Epub 2004 Aug 2. PMID 15289372
- [Background] Antonopoulos AS, Margaritis M, Shirodaria C, Antoniades C. Translating the effects of statins: from redox regulation to suppression of vascular wall inflammation. Thromb Haemost. 2012 Nov;108(5):840-8. doi: 10.1160/TH12-05-0337. Epub 2012 Aug 7. PMID 22872079
- [Background] Endres M, Laufs U, Huang Z, Nakamura T, Huang P, Moskowitz MA, Liao JK. Stroke protection by 3-hydroxy-3-methylglutaryl (HMG)-CoA reductase inhibitors mediated by endothelial nitric oxide synthase. Proc Natl Acad Sci U S A. 1998 Jul 21;95(15):8880-5. doi: 10.1073/pnas.95.15.8880. PMID 9671773
- [Background] Giannopoulos S, Katsanos AH, Tsivgoulis G, Marshall RS. Statins and cerebral hemodynamics. J Cereb Blood Flow Metab. 2012 Nov;32(11):1973-6. doi: 10.1038/jcbfm.2012.122. Epub 2012 Aug 29. PMID 22929438
- [Background] Xu G, Fitzgerald ME, Wen Z, Fain SB, Alsop DC, Carroll T, Ries ML, Rowley HA, Sager MA, Asthana S, Johnson SC, Carlsson CM. Atorvastatin therapy is associated with greater and faster cerebral hemodynamic response. Brain Imaging Behav. 2008 Jun 1;2(2):94. doi: 10.1007/s11682-007-9019-7. PMID 20157644
- [Background] De Keyser J, Steen C, Mostert JP, Koch MW. Hypoperfusion of the cerebral white matter in multiple sclerosis: possible mechanisms and pathophysiological significance. J Cereb Blood Flow Metab. 2008 Oct;28(10):1645-51. doi: 10.1038/jcbfm.2008.72. Epub 2008 Jul 2. PMID 18594554
- [Background] D'haeseleer M, Beelen R, Fierens Y, Cambron M, Vanbinst AM, Verborgh C, Demey J, De Keyser J. Cerebral hypoperfusion in multiple sclerosis is reversible and mediated by endothelin-1. Proc Natl Acad Sci U S A. 2013 Apr 2;110(14):5654-8. doi: 10.1073/pnas.1222560110. Epub 2013 Mar 18. PMID 23509249
- [Background] Paling D, Thade Petersen E, Tozer DJ, Altmann DR, Wheeler-Kingshott CA, Kapoor R, Miller DH, Golay X. Cerebral arterial bolus arrival time is prolonged in multiple sclerosis and associated with disability. J Cereb Blood Flow Metab. 2014 Jan;34(1):34-42. doi: 10.1038/jcbfm.2013.161. Epub 2013 Sep 18. PMID 24045400
- [Background] Laufs U, La Fata V, Plutzky J, Liao JK. Upregulation of endothelial nitric oxide synthase by HMG CoA reductase inhibitors. Circulation. 1998 Mar 31;97(12):1129-35. doi: 10.1161/01.cir.97.12.1129. PMID 9537338
- [Background] Mraiche F, Cena J, Das D, Vollrath B. Effects of statins on vascular function of endothelin-1. Br J Pharmacol. 2005 Mar;144(5):715-26. doi: 10.1038/sj.bjp.0706114. PMID 15678081
- [Background] Pahan K, Sheikh FG, Namboodiri AM, Singh I. Lovastatin and phenylacetate inhibit the induction of nitric oxide synthase and cytokines in rat primary astrocytes, microglia, and macrophages. J Clin Invest. 1997 Dec 1;100(11):2671-9. doi: 10.1172/JCI119812. PMID 9389730
- [Background] van der Most PJ, Dolga AM, Nijholt IM, Luiten PG, Eisel UL. Statins: mechanisms of neuroprotection. Prog Neurobiol. 2009 May;88(1):64-75. doi: 10.1016/j.pneurobio.2009.02.002. Epub 2009 Feb 21. PMID 19428962
- [Background] Schmeer C, Kretz A, Isenmann S. Statin-mediated protective effects in the central nervous system: general mechanisms and putative role of stress proteins. Restor Neurol Neurosci. 2006;24(2):79-95. PMID 16720944
- [Background] Miller E, Mrowicka M, Saluk-Juszczak J, Ireneusz M. The level of isoprostanes as a non-invasive marker for in vivo lipid peroxidation in secondary progressive multiple sclerosis. Neurochem Res. 2011 Jun;36(6):1012-6. doi: 10.1007/s11064-011-0442-1. Epub 2011 Mar 12. PMID 21399906

RESULTS

PARTICIPANT FLOW:
Groups:
- Simvastatin: Simvastatin is part of the pharmacotherapeutic group of HMG-CoA reductase inhibitors (ATC-Code: C10A A01). Simvastatin is licensed within the EU for hypercholesterolemia and cardiovascular prevention but for this trial its use will be outside its licensed indication.
  The starting dose at baseline was 40 mg of Simvastatin or placebo (one tablet) to be taken orally in the evening. This was up titrated at Visit 2 (week 4) to 80 mg (two tablets) if all safety parameters were met at Visit 2. Participants were allocated one bottle each containing 220 tablets for the duration of the study. There was therefore one drug dispensation at baseline, and the patient was reminded to up-titrate after one month at Visit 2.
- Placebo: Matched placebo taking a dummy pill (Placebo IMP: gelatine tablet with added cellulose microcrystalline).
  The starting dose at baseline for placebo was 1 tablet to be taken orally in the evening. This was up titrated at Visit 2 (week 4) to 2 tablets if all safety parameters were met at Visit 2. Participants were allocated one bottle each containing 220 tablets for the duration of the study. There was therefore one drug dispensation at baseline, and the patient was reminded to up-titrate after one month at Visit 2.
Period: Overall Study
Arm/Group | Simvastatin | Placebo
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Forty patients, including primary progressive MS and secondary progressive MS, aged 18-70 years, and presenting with an Expanded Disability Status Scale (EDSS) score 4.0-6.5 were randomly assigned (1:1) to Simvastatin 80 mg or placebo for 16 weeks.
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin | Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Forty patients, including 12 primary progressive MS and 28 secondary progressive MS, aged 18-70 years, and presenting with an Expanded Disability Status Scale (EDSS) score 4.0-6.5 were randomly assigned (1:1) to Simvastatin 80 mg or placebo for 16 weeks.
  Years | 55.30 (7.51) | 52.95 (9.48) | 54.13 (8.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 20 | 18 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 20 | 20 | 40
Multiple Sclerosis Clinical Phenotype, Categorical [Count of Participants; unit: Participants] — Clinical course at onset according to Lublin criteria
  Participants
    Primary Progressive Multiple Sclerosis | 6 | 6 | 12
    Secondary Progressive Multiple Sclerosis | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Effect on Cerebral Blood Flow in White Matter, Gray Matter, Deep White Matter, Deep Gray Matter, and Thalamus
Description: To compare patients on simvastatin or placebo using multiple linear regressions. ASL is an MRI method that allows non-invasive measurement of CBF using inversion of arterial water spins as a tracer.The aim is to explore whether subtle changes in CBF occur over time between placebo and simvastatin treated patients, including potential waning of the effects of the drug over time.
Time Frame: At week 16
Population: Mean percentage of change in CBF from baseline to visit 3 (95%CI)
Measure: Mean (95% Confidence Interval); unit: Percentage of change in CBF
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 18 | 20
Percentage of change in CBF
  White Matter | 8.55 [-1.63 to 14.77] | 5.12 [-4.52 to 14.77]
  Gray Matter | 5.78 [-2.13 to 13.69] | 2.06 [-5.43 to 9.54]
  Deep White Matter | 8.39 [-2.55 to 19.33] | 6.69 [-3.67 to 17.05]
  Deep Gray Matter | 7.33 [-1.20 to 15.85] | 2.77 [-5.07 to 10.61]
  Thalamus | 4.55 [-5.11 to 14.21] | -1.02 [-9.91 to 7.86]

2. Primary Outcome: AOSLO Measurements of Blood Flow
Description: To establish if Adaptive Optics Scanning Laser Ophthalmoscope (AOSLO) measurements of blood flow are useful correlates for cerebral blood flow measurement on and off treatment.
Time Frame: At week 16
Population: Mean percentage of change in ratio Velocity/Vessel Width from baseline to visit 3
Measure: Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 17 | 17
percentage of change | 0.87 [-15.12 to 16.86] | 5.89 [-10.11 to 21.88]

3. Secondary Outcome: MRI: ASL in White Matter, Gray Matter, Deep White Matter, Deep Gray Matter, and Thalamus
Description: To evaluate whether ASL is useful correlate for cerebral blood flow measurement on and off treatment.
Time Frame: At baseline
Population: Data are reported for ASL CBF at baseline
Measure: Mean (Standard Deviation); unit: mL/100 g/min
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 18 | 20
mL/100 g/min
  White Matter | 27.38 (8.30) | 25.89 (7.56)
  Gray Matter | 76.82 (18.02) | 70.78 (15.74)
  Deep White Matter | 24.95 (7.74) | 23.26 (7.56)
  Deep Gray Matter | 46.33 (11.95) | 44.72 (11.27)
  Thalamus | 54.96 (17.52) | 51.22 (13.75)

4. Secondary Outcome: AOSLO Blood Flow Dynamics
Description: AOSLO of retinal capillary microvessels was applied to calculate retinal perfusion and measure blood flow dynamics at the capillary level. We measured relative venous and artery blood pO2 levels near the optic nerve (central 3 disk diameters) to obtain vessel width and velocity.
Time Frame: Over 16 weeks
Population: Mean percentage of change from baseline to visit 3
Measure: Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 19 | 18
Percentage of change
  Vessel width | -3.04 [-15.93 to 9.84] | -2.64 [-14.76 to 9.48]
  Velocity | -13.40 [-25.50 to 1.29] | 5.37 [-7.10 to 17.84]

5. Secondary Outcome: MRI: Brain Atrophy
Description: To explore whether statin reduce the rate of brain atrophy, including grey matter volumes, on MRI (excluding the effect of pseudo-atrophy, which is a temporary response to the drug rather than an actual loss of tissue). The MRI images will be analysed using softwares developed at UCL to quantify the amount of brain tissue loss over time.
Time Frame: At week 16
Population: Mean prcentage of change from baseline to visit 3
Measure: Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 18 | 20
Percentage of change
  White Matter | -0.21 [-0.79 to 0.36] | 0.14 [-1.17 to 0.46]
  Gray Matter | -0.32 [-0.74 to 0.09] | -0.19 [-0.58 to 0.20]
  Cortical Gray Matter | -0.32 [-0.75 to 0.10] | -0.20 [-0.60 to 0.20]
  Hippocampus | -0.51 [-1.11 to 0.09] | -0.44 [-1.00 to 0.13]
  Thalamus | -0.25 [-0.91 to 0.42] | -0.04 [-0.67 to 0.59]
  Pallidum | 0.15 [-0.79 to 1.09] | -0.68 [-1.57 to .021]
  Putamen | -0.30 [-0.80 to 0.21] | -0.85 [-1.34 to -0.38]
  Ventral diencephalon | 0.09 [-0.48 to 0.66] | -0.85 [-1.39 to 0.32]

6. Secondary Outcome: MRI: Diffusion Tensor Imaging (DTI)
Description: Diffusion weighted imaging (DWI) is an MR imaging technique based upon the measurement of the random Brownian motion of water within a voxel of tissue. This technique has been used to analyse the microstructure of neuronal tissue in particular myelin and axonal integrity.
Time Frame: At week 16
Population: Mean percentage of change from baseline to visit 3. Data are reported for white matter
Measure: Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 18 | 19
Percentage of change
  Fractional anisotropy (FA) | -0.01 [-0.95 to 0.92] | -0.22 [-1.14 to 0.69]
  Mean diffusivity (MD) | 1.13 [0.01 to 2.26] | 0.31 [-0.78 to 1.40]

7. Secondary Outcome: MRI: Neurite Density and Orientation Dispersion Imaging
Description: To assess changes in axonal parameters, such as fiber orientation dispersion and axonal densities occurring over time using NODDI, an advanced MRI technique that reflects the microstructural complexity of dendrites and axons in vivo.
Time Frame: At week 16
Population: Mean percentage of change from baseline to visit 3. Data are reported for white matter
Measure: Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 18 | 19
Percentage of change
  Intra-neurite volume fraction | -1.27 [-2.58 to 0.04] | -0.48 [-1.75 to 0.79]
  Isotropic volume fraction | 2.45 [-0.58 to 5.47] | -0.12 [-3.06 to 2.83]

8. Secondary Outcome: MRI: MTV
Description: Macromolecular tissue volume (MTV) is a method of myelin mapping to determine the role of myelin loss or changes in progressive MS. With the macromolecular volume being made up of 50% myelin, we are able to use an in-house analysis pipeline to calculate the MTV - a surrogate marker of brain myelin volume. This metric, alongside diffusion weighted imaging will provide micro-structural detail into the cross-sectional and longitudinal changes occurring in the brain parenchyma of people with progressive MS.
Time Frame: At week 16
Population: Mean percentage of change from baseline to visit 3
Measure: Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 18 | 19
Percentage of change
  Cortical Gray Matter | 3.65 [-8.29 to 15.59] | 7.30 [-4.30 to 18.89]
  Deep Gray Matter | -2.27 [-7.31 to 2.77] | 1.89 [-3.01 to 6.79]
  Normal-Appearing White Matter | -0.68 [-4.72 to 3.36] | 1.77 [-2.15 to 5.70]
  Brainstem | -1.69 [-7.22 to 3.83] | 1.71 [-3.65 to 7.08]
  Lesions | -2.12 [-7.79 to 3.56] | 2.66 [-2.86 to 8.17]

9. Secondary Outcome: OCT-A: Retinal Nerve Fibre Layer
Description: Inner retinal thickness will be measured using optical coherence tomography (OCT). OCT is a method of retinal imaging which is non-invasive and involves the patient holding their head still and staring at a dim light while imaging takes place. Peripapillary retinal nerve fibre layer (pRNFL) thickness is a strong candidate as a biomarker of axonal degeneration in MS.
Time Frame: At week 16
Population: Mean percentage of change from baseline to visit 3
Measure: Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 16 | 18
Percentage of change | 2.28 [-0.08 to 4.64] | -0.29 [-2.52 to 1.93]

10. Secondary Outcome: OCT-A: Vessel Density
Description: OCT-A images will be processed to produce quantitative data of perfusion indices. Vessel density (VD) is defined as the "percentage area occupied by vessels in the segmented area.
Time Frame: At week 16
Population: Mean percentage of change from baseline to visit 3
Measure: Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 16 | 19
Percentage of change | 7.59 [-11.12 to 26.30] | 15.15 [-1.97 to 32.26]

11. Secondary Outcome: Clinical Outcome: EDSS
Description: To examine the clinical effect of simvastatin treatment as reported by the clinician. Clinician observed expanded disability status score (EDSS) is a method of quantifying disability in MS and records changes in disability over time. The EDSS scale ranges from 0 (no disability) to 10 (death due to MS) in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist and encompasses pyramidal, cerebellar, brainstem, sensory, bowel/bladder function in addition to visual, cerebral and other functions. Changes in score (including no changes) will be recorded to determine progression of disability.
Time Frame: At week 16
Population: Mean change from baseline to visit 3
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 18 | 20
units on a scale | -0.19 [-0.46 to 0.08] | 0.04 [-0.21 to 0.30]

12. Secondary Outcome: Clinical Outcomes: MSFC: 25 Foot Timed Walk
Description: To examine the clinical effect of simvastatin treatment as reported by the clinician . Multiple Sclerosis Function Composite (MSFC) includes the 25 foot timed foot walk (25TFW), which involves marking a 25-foot distance in an unobstructed hallway; an assistive device (if needed) may be used by the participant and recorded. Their speed is then timed up to a time limit of 3 mins in both directions. Changes in scores will be recorded over the time-points described.
Time Frame: At week 16
Population: Mean change from baseline to visit 3
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 18 | 20
Seconds | 0.74 [-6.94 to 8.41] | 2.37 [-4.90 to 9.64]

13. Secondary Outcome: Clinical Outcomes: MSFC: 9 Hole Peg Test
Description: To examine the clinical effect of simvastatin treatment as reported by the clinician. Multiple Sclerosis Function Composite (MSFC) includes the 9 hole peg test (9HPT). The 9-HPT is a quantitative measure of upper extremity (arm and hand) function. Both the dominant and non-dominant hands are tested twice (two consecutive trials of the dominant hand, followed immediately by two consecutive trials of the non-dominant hand). It is important that the 9-HPT be administered on a solid table (not a rolling hospital bedside table) and that the 9-HPT apparatus be anchored (e.g., with Dycem). The pegs are selected one at a time, using one hand only, and put into the holes as quickly as possible in any order until all the holes are filled. Then, without pausing, the pegs are removed one at a time and returned to the container. This is timed and recorded at the time-points described.
Time Frame: At week 16
Population: Mean change from baseline to visit 3
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 18 | 20
Seconds
  Dominant hand | -0.77 [-13.63 to 12.09] | 4.51 [-7.65 to 16.68]
  Non-dominant hand | 0.78 [-7.66 to 9.22] | -0.10 [-8.10 to 7.89]

14. Secondary Outcome: Clinical Outcomes: SDMT
Description: Symbol Digit Modalities Test (SDMT) is measure of cognitive impairment. The subject is asked to match single digits to symbols using a key as a guide that pairs the numbers to the symbols. They are presented with a page headed by a key that pairs the single digits 1-9 with nine symbols and they then write or orally report their responses in a scoring form. It can be administered in oral and written form and is timed and guided by a trained examiner ie. suitably qualified member of the research team. Changes in scores were recorded over the time-points described. Scores range from 0 to 110, with higher scores indicating better cognitive functioning.
Time Frame: At week 16
Population: Mean change from baseline to visit 3.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 18 | 20
Units on a scale | -2.34 [-5.94 to 1.25] | 0.01 [-3.40 to 3.42]

15. Secondary Outcome: Clinical Outcomes: Frontal Executive Functioning: FAB
Description: Frontal Assessment Battery (FAB). The FAB is a brief tool that can be used at the bedside or in a clinic setting to assist in discriminating between dementias with a frontal dysexecutive phenotype and dementia of Alzheimer"s Type (DAT). The FAB has validity in distinguishing Fronto-temporal type dementia from DAT in mildly demented patients (MMSE > 24). Total score is from a maximum of 18, higher scores indicating better performance. Changes in scores were recorded over the time-points described. The FAB evaluates executive functions through six subtests, including conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy. Each subtest is scored from 0 to 3, yielding a total score range of 0 to 18. Higher scores indicate better executive functioning. The total score is calculated by summing the six subtest scores.
Time Frame: At week 20
Population: Mean change from baseline to visit 4
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 19 | 19
Units on a scale | 0.38 [-0.24 to 1.00] | 0.40 [-0.22 to 1.03]

16. Secondary Outcome: Patient-Reported Outcomes: MSIS-29v2 Questionnaires.
Description: To examine the clinical effect of simvastatin treatment as reported by patient reported outcome measures. Patient reported multiple sclerosis impact scale version 2 (MSIS-29v2) is a self-administered questionnaire covering 29 items that asks to what degree MS has impacted the person physically and mentally over the past two weeks. It consists of 29 items divided into two subscales: Physical Impact (20 items; score range: 20-100) and Psychological Impact (9 items; score range: 9-45). Each item is rated on a 5-point Likert scale. Higher scores reflect a greater negative impact of MS on the individual's quality of life.
Time Frame: At week 16
Population: Mean change in total score from baseline to visit 3. The FAB evaluates executive functions through six subtests, including conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy. Each subtest is scored from 0 to 3, yielding a total score range of 0 to 18. Higher scores indicate better executive functioning. The total score is calculated by summing the six subtest scores.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 18 | 20
Units on a scale
  Physical impact | 1.08 [-4.53 to 6.69] | -5.09 [-10.39 to 0.20]
  Psychological impact | 1.54 [-5.11 to 8.19] | 1.81 [-4.48 to 8.10]

17. Secondary Outcome: Patient-Reported Outcomes: MSWT-12V2 Questionnaires.
Description: Patient reported Multiple Sclerosis Walking Test version 2 (MSWT-12V2) is a 12 item self-administered questionnaire that measures walking performance over the previous two weeks. Each items is summed to generate a total score which is then transformed to a scale ranging from 0 to 100. Higher scores indicate greater impact on walking. Changes in scores will be recorded over the time-points described.
Time Frame: At week 16
Population: Mean change from baseline to visit 3
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 17 | 19
Units on a scale | 1.43 [-3.46 to 6.31] | 3.15 [-1.46 to 7.77]

18. Secondary Outcome: Health Economic Outcomes: EQ5D5L
Description: The EuroQol Health-Related Quality of Life (EQ-5D-5L) is a standardized instrument for assessing health-related quality of life across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is rated on a five-level scale, ranging from 1 (no problems) to 5 (extreme problems). The EQ-5D-5L also includes a visual analogue scale (VAS), on which individuals rate their overall health from 0 (worst imaginable health state) to 100 (best imaginable health state). Results are reported as the mean change in domain scores and VAS ratings from baseline to Visit 3.
Time Frame: At week 16
Population: Mean change from baseline to visit 3
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 18 | 20
Units on a scale
  Mobility | 0.11 [-0.09 to 0.32] | 0.20 [0.001 to 0.39]
  Self-care | -0.09 [-0.39 to 0.20] | -0.07 [-0.35 to 0.21]
  Usual activities | 0.15 [-0.18 to 0.49] | 0.11 [-0.21 to 0.43]
  Pain/discomfort | 0.25 [-0.06 to 0.55] | 0.18 [-0.11 to 0.46]
  Anxiety/depression | -0.08 [-0.42 to 0.27] | 0.07 [-0.26 to 0.39]
  VAS | 4.20 [-1.41 to 9.81] | 2.07 [-3.25 to 7.39]

19. Other Pre Specified Outcome: Exploratory Outcomes: Immune Parameters, and Biomarkers.
Description: Blood samples from these patients will be taken at baseline and at weeks 4, 16 and 20 to investigate the effect of statins on vascular leakage and free radical damage. Biomarkers will be determined as follows: (i) For RNA/DNA oxidative damage serum levels of 8-hydroxyguanosine (8-OHG)/8-hydroxydeoxyguanosine (8-OHdG); (ii) Protein oxidative damage will be determined by assaying plasma proteins for nitrotyrosine and carbonyl content; and (iii) Detection of lipid oxidative damage by assaying for the advanced lipid peroxidation end products 4-hydroxynonenal (4-HNE or HNE), malondialdehyde (MDA), 8-iso-prostaglandin F2α and thiobarbituric acid reactive substances (TBARS) (Miller et al., 2012).
Time Frame: At week 4
Population: Mean percentage of change from baseline to visit 2
Measure: Mean (95% Confidence Interval); unit: Percentage of change
Arm/Group | Simvastatin | Placebo
Number analyzed (Participants) | 15 | 18
Percentage of change
  Nos. Lymph events gated | -381.57 [-1151.38 to 388.24] | -280.97 [-958.49 to 396.55]
  Nos. CD3+T cell events gated | 196.26 [-1035.94 to 1428.46] | 286.48 [-798.13 to 1371.09]
  CD4+ T cells | -113.84 [-238.98 to 11.30] | 13.73 [-99.59 to 127.04]
  CD8+ T cells | -344.68 [-615.56 to -73.79] | -209.93 [-463.84 to 43.98]
  B cells | -74.50 [-464.45 to 315.45] | -253.57 [-606.90 to 99.74]
  CD8+ non-T cells | -110.50 [-209.31 to 11.69] | -41.85 [-137.44 to 53.74]
  CD4+ IFN+ (Th1) cells | -37.60 [-672.04 to 596.84] | 165.81 [-425.07 to 756.68]
  CD4+ IL17+ (Th17) cells | -138.72 [-313.51 to 36.06] | -71.45 [-240.23 to 97.32]
  8OH | -24.40 [-53.26 to 4.46] | 26.69 [-0.40 to 53.77]
  Nitro | 59.14 [10.40 to 107.87] | 66.60 [25.78 to 107.42]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a period of 3 years and 4 months, and more specifically, from June June 2019 (the enrollment date of the first patient) to 12th October 2022 (one month after the final visit of the last patient). Adverse event data were collected for each participant from baseline through one month after their final study visit, resulting in an individual assessment period of approximately 24 weeks per participant, depending on their enrollment and visit schedule.
Description: Adverse Event (AE): Any untoward medical occurrence in a patient or clinical trial participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment.
  Serious Adverse Event (SAE), Serious Adverse Reaction (SAR) or Unexpected Serious Adverse Reaction: Any adverse event, adverse reaction or unexpected adverse reaction, respectively, that: results in death
Arm/Group | Simvastatin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 6/20 | 11/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Simvastatin (N=20) | Placebo (N=20)
Increased TSH (Endocrine disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flu (General disorders) | 0 (0) | 1 (1)
Increased ALT and/or AST (Hepatobiliary disorders) | 3 (3) | 0 (0)
Dental infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Bone fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Muscle pain and stiffness (Musculoskeletal and connective tissue disorders) | 2 (3) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Increased CK (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Movement disorder (Nervous system disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Numbness (Nervous system disorders) | 0 (0) | 2 (2)
Fatigue (General disorders) | 1 (1) | 1 (1)
Speech difficulties (Nervous system disorders) | 0 (0) | 1 (1)
Brain fog (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03896217/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT03896217/SAP_001.pdf
  • Informed Consent Form (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/17/NCT03896217/ICF_002.pdf